CLINICAL TRIAL: NCT01785212
Title: The Influence of Two Different Hepatectomy Methods on Transection Speed and Chemokine Release From the Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Klaus Kaczirek, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 1.0
Record Dates: First submitted 2013-01-23; First posted 2013-02-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Liver Neoplasms; Liver Metastasis; Liver Hemangioma; Echinococcosis, Hepatic
MeSH Terms: conditions — Liver Neoplasms; Echinococcosis, Hepatic | interventions — Surgical Staplers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stapler-hepatectomy (Other): The liver parenchyma is crushed with a Pean clamp and subsequently divided using Covidien Endo-Gia™ Ultra Handle Short Staplers and Endo Gia™ TRI staple 60 mm or 45 mm AVM/AMT loading units (Covidien). Hepatic veins and portal pedicles clamped and suture ligated.
  Interventions: Device: Stapler
- CUSA-hepatectomy (Other): The liver parenchyma is divided along the transection line by CUSA (Cavitron ultrasonic aspirator; Valleylab, Boulder, CO) and bipolar forceps in a two surgeon technique. Vessels of less than 2 mm in diameter are coagulated with bipolar forceps. The remaining vessels are clipped or ligated. Hepatic veins and portal pedicles clamped and suture ligated.
  Interventions: Device: CUSA (Cavitron ultrasonic aspirator; Valleylab, Boulder, CO)

INTERVENTIONS:
Device: Stapler — stapler hepatectomy
  Other Names: Covidien Endo-Gia™ Ultra Handle Short Staplers(Covidien)
  Arms: Stapler-hepatectomy
Device: CUSA (Cavitron ultrasonic aspirator; Valleylab, Boulder, CO) — CUSA is a well established device used for hepatic resection using ultrasound
  Arms: CUSA-hepatectomy

SUMMARY:
The CUSA (cavitron ultrasound surgical aspirator) is the method of choice for hepatic resection in our center. Recently a stapler-hepatectomy methods has been developed and approved for liver surgery using Covidien Endo-Gia stapler. The potential benefit of this method is a potential shorter transection time compared to the CUSA technique. Thus the investigators will perform a randomized controlled trial including 20 patients in the stapler-group and 20 patients in the CUSA control group. Primary endpoint will be transection speed. Secondary endpoints will be peri-operative (d-1, d0, d1, d3) cytokines concentration, T cell subsets, blood loss, morbidity, and a cost analysis.

DETAILED DESCRIPTION:
Many different techniques of parenchymal transection are used in hepatic surgery. In a systematic review, there were no significant differences in morbidity (including bile leak), mortality, routine markers of liver parenchymal injury or dysfunction and length of hospital stay irrespective of the method used for parenchymal transection. This Cochrane review analyzed studies comparing the following transection devices: CUSA (cavitron ultrasound surgical aspirator) versus clamp-crush (two trials); radiofrequency dissecting sealer versus clamp-crush (two trials); sharp dissection versus clamp-crush technique (one trial); and hydrojet versus CUSA (one trial). The clamp-crush technique appeared to have the lowest blood loss and lowest transfusion requirements compared to the other techniques.

However, even in specialized centers morbidity and mortality rates of hepatic resections are still in the range of 45% and 3% respectively and uncertainty persists regarding the optimal technique of transection. Local experience seems to be the most important factor for the choice of the transection method. An innovative technique is stapler hepatectomy using Covidien Endo-Gia™ Ultra Handle Short Staplers and Endo Gia™ TRI staple 60mm or 45 mm AVM/AMT loading units (Covidien). A randomized controlled trial (CRUNSH trial) to evaluate the intraoperative blood loss of stapler hepatectomy compared to the clamp-crushing technique is currently under way.

The CUSA technique is well established in many centers including ours with excellent morbidity and mortality rates. However, it has been shown that CUSA has a longer transection speed than the clamp-crush technique (with vascular occlusion). The investigators of the CRUNSH trial hypothesize that stapler hepatectomy technique might also be comparable or more favorable to clamp-crushing regarding transection time with the advantage of avoiding vascular occlusion. Therefore stapler hepatectomy should also be faster than CUSA.

It has been shown that the release of cytokines, chemokines, and stress hormones correlates with postoperative infection and organ dysfunction. Chemokines are critically involved in the process of leukocyte recruitment and activation in the liver. Major surgery causes inflammation reflected in the production of pro-inflammatory cytokines. In various studies IL-6, for instance, was a valid predictor for post-operative sepsis, complications or mortality. Besides, the levels of these cytokines are expected to correlate with the degree of surgical trauma. Therefore differences in cytokine levels between the two study groups will be assessed, including pro- (INF-γ, IL-1β, IL-5, IL-6, IL12p70, TNFα) and anti-inflammatory (IL-4, IL-10, IL-13) cytokines.

Monocyte chemotactic protein-1 (MCP-1) production is elevated in Kupffer cells following ischemia / reperfusion in response to free radicals and neutrophil elastase, as well as in animal oxidative liver injury models (e.g. carbon tetrachloride) Macrophage inflammatory protein-3-alpha (MIP3-alpha) is constitutively expressed in the liver. It is strongly chemotactic for cytokine-stimulated neutrophils, immature dendritic cells and memory/effector T and B lymphocytes by utilizing chemokine receptor (CCR) 6.

sCD163 (soluble haemoglobin scavenger receptor) is a novel marker of activated macrophages, like neopterin it can be determined in serum or plasma.

The effect of the transection speed in respect to chemokine release has never been investigated. The investigators hypothesize that a shorter transection time leads to a reduced release of these molecules potentially resulting in improved postoperative outcome.

Additionally the interaction between adaptive and innate immunity plays a significant role in liver ischemia-reperfusion (I/R) injury. Notably, activation of T cells in the absence of TCR ligation seems to be a predominant factor in the initial phase of I/R injury. Therefore as a pilot study, peripheral T cell subsets (including naïve T cells, effector and central memory T cells, regulatory T cells, early activated T cells) will be determined by flow cytometry in a subgroup of study patients (i.e. patients undergoing hepatic resection for other than oncological reasons).

The supposedly slower technique of CUSA resection shall therefore be compared with the novel technique of stapler hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective major hepatic resection at the Department of General Surgery, Medical University of Vienna
* Stapler hepatectomy and CUSA resection feasible based on preoperative imaging
* Age equal or greater than 18 years
* Informed consent

Exclusion Criteria:

* Minor hepatectomy
* Hepatitis B, Hepatitis C, HIV infection, autoimmune disease
* Inflammatory conditions of the bowel such as Crohn's Disease
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
transection speed | during surgery
  The transection time will be recorded by the anesthesiological team during surgery. The transection phase starts with opening the liver parenchyma after the transection line has been marked by electrocautery. It ends after complete division of the liver parenchyma. The cut surface of the resected liver will be photographed together with a 4 cm² reference scale in an exact 90° angle. The area of the liver transection surface will be calculated in cm² by setting the measured pixels of the cut surface in relation to the reference scale using Adobe Photoshop. The transection speed will expressed in cm²/min

SECONDARY OUTCOMES:
Perioperative cytokine concentrations | day -1, d0, d1, d3
Intraoperative blood loss in ml | during surgery
Postoperative laboratory markers of liver damage | first week after surgery
  Postoperative routine laboratory markers of liver damage (aspartate aminotransferase (AST), alanine aminotransferase (ALT)), and markers of liver function (bilirubin, prothrombin time) measured on first and third postoperative day
Morbidity and Mortality | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Perioperative T-cell subsets | Day -1, 0, 1, 3

OTHER OUTCOMES:
Costs and health economics | participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kaczirek, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Dept. of Surgery/Div. of General Surgery Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Gurusamy KS, Pamecha V, Sharma D, Davidson BR. Techniques for liver parenchymal transection in liver resection. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD006880. doi: 10.1002/14651858.CD006880.pub2. PMID 19160307
- [Background] Jarnagin WR, Gonen M, Fong Y, DeMatteo RP, Ben-Porat L, Little S, Corvera C, Weber S, Blumgart LH. Improvement in perioperative outcome after hepatic resection: analysis of 1,803 consecutive cases over the past decade. Ann Surg. 2002 Oct;236(4):397-406; discussion 406-7. doi: 10.1097/01.SLA.0000029003.66466.B3. PMID 12368667
- [Background] Rahbari NN, Elbers H, Koch M, Bruckner T, Vogler P, Striebel F, Schemmer P, Mehrabi A, Buchler MW, Weitz J. Clamp-crushing versus stapler hepatectomy for transection of the parenchyma in elective hepatic resection (CRUNSH)--a randomized controlled trial (NCT01049607). BMC Surg. 2011 Sep 4;11:22. doi: 10.1186/1471-2482-11-22. PMID 21888669
- [Background] Tamandl D, Gruenberger B, Herberger B, Kaczirek K, Gruenberger T. Surgery after neoadjuvant chemotherapy for colorectal liver metastases is safe and feasible in elderly patients. J Surg Oncol. 2009 Oct 1;100(5):364-71. doi: 10.1002/jso.21259. PMID 19235181
- [Background] Tamandl D, Gruenberger B, Klinger M, Herberger B, Kaczirek K, Fleischmann E, Gruenberger T. Liver resection remains a safe procedure after neoadjuvant chemotherapy including bevacizumab: a case-controlled study. Ann Surg. 2010 Jul;252(1):124-30. doi: 10.1097/SLA.0b013e3181deb67f. PMID 20562613
- [Background] Kimura F, Shimizu H, Yoshidome H, Ohtsuka M, Kato A, Yoshitomi H, Nozawa S, Furukawa K, Mitsuhashi N, Sawada S, Takeuchi D, Ambiru S, Miyazaki M. Circulating cytokines, chemokines, and stress hormones are increased in patients with organ dysfunction following liver resection. J Surg Res. 2006 Jun 15;133(2):102-12. doi: 10.1016/j.jss.2005.10.025. Epub 2006 Jan 4. PMID 16386757
- [Background] Yamauchi H, Kobayashi E, Yoshida T, Kiyozaki H, Hozumi Y, Kohiyama R, Suminaga Y, Sakurabayashi I, Fujimura A, Miyata M. Changes in immune-endocrine response after surgery. Cytokine. 1998 Jul;10(7):549-54. doi: 10.1006/cyto.1997.0322. PMID 9702420
- [Background] Cruickshank AM, Fraser WD, Burns HJ, Van Damme J, Shenkin A. Response of serum interleukin-6 in patients undergoing elective surgery of varying severity. Clin Sci (Lond). 1990 Aug;79(2):161-5. doi: 10.1042/cs0790161. PMID 2167805
- [Background] Baigrie RJ, Lamont PM, Kwiatkowski D, Dallman MJ, Morris PJ. Systemic cytokine response after major surgery. Br J Surg. 1992 Aug;79(8):757-60. doi: 10.1002/bjs.1800790813. PMID 1393463
- [Background] Mokart D, Merlin M, Sannini A, Brun JP, Delpero JR, Houvenaeghel G, Moutardier V, Blache JL. Procalcitonin, interleukin 6 and systemic inflammatory response syndrome (SIRS): early markers of postoperative sepsis after major surgery. Br J Anaesth. 2005 Jun;94(6):767-73. doi: 10.1093/bja/aei143. Epub 2005 Apr 22. PMID 15849208
- [Background] Jawa RS, Anillo S, Huntoon K, Baumann H, Kulaylat M. Interleukin-6 in surgery, trauma, and critical care part II: clinical implications. J Intensive Care Med. 2011 Mar-Apr;26(2):73-87. doi: 10.1177/0885066610384188. PMID 21464062
- [Background] Zhai Y, Busuttil RW, Kupiec-Weglinski JW. Liver ischemia and reperfusion injury: new insights into mechanisms of innate-adaptive immune-mediated tissue inflammation. Am J Transplant. 2011 Aug;11(8):1563-9. doi: 10.1111/j.1600-6143.2011.03579.x. Epub 2011 Jun 10. PMID 21668640
- [Background] Caldwell CC, Tschoep J, Lentsch AB. Lymphocyte function during hepatic ischemia/reperfusion injury. J Leukoc Biol. 2007 Sep;82(3):457-64. doi: 10.1189/jlb.0107062. Epub 2007 Apr 30. PMID 17470532
- [Derived] Schwarz C, Klaus DA, Tudor B, Fleischmann E, Wekerle T, Roth G, Bodingbauer M, Kaczirek K. Transection Speed and Impact on Perioperative Inflammatory Response - A Randomized Controlled Trial Comparing Stapler Hepatectomy and CUSA Resection. PLoS One. 2015 Oct 9;10(10):e0140314. doi: 10.1371/journal.pone.0140314. eCollection 2015. PMID 26452162